CLINICAL TRIAL: NCT04805814
Title: The Clinical Utility Of Cardiac Magnetic Resonance Imaging in Patients With Angina But No Obstructive Coronary Disease (CorCMR): A Diagnostic Study And Nested Randomised Trial
Brief Title: Coronary Microvascular Angina Cardiac Magnetic Resonance Imaging (CorCMR) Trial
Acronym: CorCMR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: University of Glasgow (Other); British Heart Foundation (Other); Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Principal Investigator, Colin Berry, Chief Investigator, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 281128
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Microvascular Angina; Angina Pectoris; Angina, Stable; Non-Obstructive Coronary Atherosclerosis; Small Vessel Cerebrovascular Disease; Coronary Artery Disease
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris; Angina, Stable; Cerebral Small Vessel Diseases; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): All randomised participants will receive stratified medicine. The subjects will undergo stress perfusion CMR as an adjunct to invasive coronary angiography. The CMR results will be disclosed to the clinician to clarify endotypes and re-evaluate the clinical diagnosis. Linked guideline-directed medical therapy and lifestyle measures will be recommended based on the endotype. The patient and clinicians responsible for downstream care will not be informed of the randomised group but they will be informed of the endotype and linked treatment plan, in the same way as in the Standard Care control group. They will be blinded to the allocated study arm and CMR findings.
  Interventions: Diagnostic Test: CMR results disclosed
- Standard Care Group (Sham Comparator): All randomised participants in this arm will receive standard angiography-guided care. The endotype will be determined based on the angiogram and all of the available clinical information. The participants in this group will also undergo stress perfusion CMR but the results will not be disclosed. Management of the patient is as per standard of care, with therapy linked to the diagnosis (endotype). The patient and clinicians responsible for downstream care will not be informed of the randomised group but they will be informed of the endotype and linked treatment plan in the same way as in the Intervention Group. They will be blinded to the allocated study arm and CMR findings.
  Interventions: Diagnostic Test: CMR performed but results not disclosed

INTERVENTIONS:
Diagnostic Test: CMR results disclosed — The results of the CMR are disclosed, and used to guide management
  Arms: Intervention Group
Diagnostic Test: CMR performed but results not disclosed — The results of the CMR are not disclosed, and management is angiography-guided
  Arms: Standard Care Group

SUMMARY:
Anginal symptoms due to ischaemia with no obstructive coronary arteries (INOCA) is a common clinical problem, however, diagnosis and onward management is heterogeneous, and prognosis is affected. Recent advances in quantifying myocardial blood flow using stress perfusion cardiac magnetic resonance imaging (CMR) has potential for accurate detection coronary microvascular dysfunction.

The CorCMR diagnostic study involves stress perfusion CMR in patients with suspected INOCA to clarify the prevalence of subgroups of patients with underlying problems, such as microvascular disease or undisclosed obstructive coronary artery disease, that might explain their anginal symptoms.

A nested, prospective, randomised, controlled, double-blind trial will determine whether stratified medical therapy guided by the results of the stress perfusion CMR improves symptoms, well-being, cardiovascular risk and health and economic outcomes.

DETAILED DESCRIPTION:
Background:

There are approximately 2 million men and women living with angina in the UK. In 2014, there were ~247,000 coronary angiograms performed, mostly for the investigation of known or suspected angina. However, obstructive CAD is detected in only 1 in 2 patients. The explanation for the cause(s) of the chest pain are often unclear. Microvascular or vasospastic angina may be one explanation.

Adjunctive tests of coronary artery function to diagnose these problems are rarely used during coronary angiography in the NHS, meaning that patient management may be empirical and heterogeneous. The lack of adoption of these novel tests in the NHS reflects key gaps in the clinical evidence. It is these gaps, coupled with the increasing adoption of anatomical coronary artery imaging with CT coronary angiography (CTCA), which stimulate this research. In recent large clinical trials, CT coronary angiography has been shown not to reduce the rate of invasive angiography. In fact, compared to standard care based on stress testing, CTCA is associated with less improvement in anginal symptoms and in quality of life (PUBMED ID: 28246175). Anatomical tests, such as CTCA and invasive angiography, do not provide information on myocardial blood flow. New evidence that addresses these gaps might inform therapy development and future trials.

Current gaps in evidence and guidelines point to a problem of unmet need in the NHS care pathway. Stress perfusion CMR has potential diagnostic value for microvascular disease, but whether it might discriminate clinical endotypes in a relatively unselected population of patients in daily practice, is uncertain. Further, access to stress perfusion CMR varies widely not least because evidence from randomised trials supporting clinical and economic benefits from a CMR-guided approach is lacking. CorCMR is a clinical strategy trial that is designed to address this evidence gap.

Hypothesis:

In patients with angina in whom obstructive disease in the epicardial coronary arteries has been ruled out by coronary angiography ± FFR, stress perfusion CMR will reclassify the diagnosis leading to changes in treatment (start or stop therapy), improvements in health and economic outcomes, as compared to decisions based standard care (CMR not disclosed).

Design:

We propose that an observational, diagnostic study involving stress CMR will provide information on the prevalence of microvascular disease in a population with anginal symptoms potentially attributable to myocardial ischaemia with no obstructive coronary arteries (INOCA). Each diagnosis is linked to a guideline-directed treatment plan.The potential value of this strategy can only be confirmed if it is associated with patient benefits, which is why we propose a nested, randomised, controlled, double-blind trial of routine disclosure of stress perfusion CMR vs. angiography-guided management

Methods:

Patients undergoing invasive coronary angiography for the investigation of known or suspected angina and who do not have either structural heart disease or a systemic health problem that would explain those symptoms will be invited to participate. Written informed consent is required for participation. Eligibility is further confirmed at the time of the coronary angiogram by exclusion of obstructive (stenosis >70% in a single segment or 50 - 70% in 2 adjacent segments in an artery >2.5 mm, or FFR ≤0.80) coronary artery disease (CAD). Angina symptoms will be confirmed by the completion of validated questionnaires and patients will be invited to attend for a stress perfusion CMR within 3 months of the original coronary angiogram.

On arrival for the CMR, patients will be randomised (1:1) to either the intervention (CMR guided, results disclosed) or blinded control group (CMR undertaken but results not disclosed, standard of care) group.

Trial participants will be blinded to treatment group. The clinicians responsible for on-going care will also be blinded. The design is therefore 'double-blind'. Following the CMR, patients and clinicians will be advised of the diagnosis (endotype) but not the randomised group. The endotype will be informed by the CMR in the intervention group but not in the control group (CMR results not disclosed, angiography-guided). Medical therapy and lifestyle measures are linked to the endotype and informed by contemporary practice guidelines. Therefore, optimal guideline-directed medical care according to the endotype is intended to be the same, regardless of the group allocation.

The sample size is 280 randomised participants. The minimum follow-up duration is 12 months from the last participant recruitment. Follow-up will continued in the longer term including, where feasible, electronic case record linkage.

The primary outcome of the diagnostic study is the reclassification of the initial diagnosis based on findings from the cardiac MRI scan. The primary outcome of the nested randomised trial is the within-subject change at 6 months from baseline for the domains of the Seattle Angina Questionnaire.

Secondary outcomes include other Patient Reported Outcome Measures (PROMS) to describe other aspects of health and wellbeing. These include EQ-5D-5L, Illness perception (Brief IPQ), Treatment satisfaction (TSQM), Duke Activity Status Index (DASI), the International Physical Activity Questionnaire (IPAQ-SF) short-form and a pain questionnaire.

There is preliminary evidence that small vessel disease can be a systemic problem affecting different organs. Whether small vessel disease in the heart might associate with small vessel disease in the brain or retina is unknown. In the CorMicA pilot study, studies of small vessels isolated from biopsies found evidence of endothelial dysfunction and increased responsiveness of the blood vessels to naturally-occurring, constriction-inducing peptides such as endothelin and thromboxane. For these reasons, we plan heart-brain-retina and peripheral vascular substudies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Symptoms of angina or angina-equivalent informed by the Rose Angina questionnaire.
3. Coronary angiography ≤3 months with a plan for medical management.

Exclusion Criteria:

1. Obstructive coronary artery disease i.e. a stenosis >70% in a single segment or 50 - 70% in 2 adjacent segments in an artery >2.5 mm, or FFR ≤0.80.
2. Coronary revascularization by percutaneous coronary intervention or coronary artery bypass graft surgery following the index angiogram.
3. Prior coronary artery bypass surgery
4. A diagnosis that would explain the angina e.g. anaemia, aortic stenosis, hypertrophic cardiomyopathy,
5. Contra-indication to contrast-enhanced CMR e.g. eGFR < 30mL/min/1.73m2.
6. Contra-indication to intravenous adenosine, i.e. severe asthma; long QT syndrome; second- or third-degree AV block and sick sinus syndrome.
7. Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Reclassification of the initial diagnosis | Day 1
  The reclassification of the initial diagnosis based on invasive management following multi-parametric stress perfusion CMR. The diagnostic groups (endotypes) are:
  1. Anginal symptoms with a myocardial perfusion defect indicative of obstructive CAD;
  2. Anginal symptoms associated with a myocardial perfusion defect indicative of microvascular disease;
  3. Vasospastic angina;
  4. Incidental finding that is actionable e.g. aortic stenosis, cardiomyopathy, lung cancer; or
  5. No clinically significant finding or normal.
Seattle Angina Questionnaire (SAQ) Summary Score | 6 months
  The 7-item version of the SAQ reflects the frequency of angina (SAQ Angina Frequency score) and the disease-specific effect of angina on patients' physical function (SAQ Physical Limitation score) and quality of life (Quality of Life score) over the previous 4 weeks; these scores are averaged to obtain the SAQ Summary score, which is an overall measure of patients' stable ischaemic heart disease-specific health status. SAQ scores range from 0 to 100, with higher scores indicating less frequent angina, improved function, and better quality of life.

SECONDARY OUTCOMES:
Compliance with the protocol | 0-36 months
  Assess feasibility of the clinical strategy by measuring compliance with the protocol and, specifically, rate of enrolment, % of patients who drop-out, % of patients who complete the diagnostic MRI protocol.
Integrity of blinding in the Radiology Department and during follow-up | 0-36 months
  Assess the integrity and feasibility of blinding by administering patient and clinician questionnaires to determine if both groups have been successfully blinded
Diagnostic utility | 0-36 months
  To assess % of patients with a change in diagnosis following disclosure of the cardiac MRI results, and relatedly, the level of certainty reported by the physicians for the diagnosis (diagnostic utility). This will be assessed by a questionnaire completed by the clinician before the MRI, and then again after the MRI results are disclosed.
Clinical Utility | 0-36 months
  To assess impact of disclosure of the cardiac MRI results on clinical management (including treatment and investigations). This will be measured by asking clinicians to complete a questionnaire on ongoing clinical management following disclosure of the MRI result
Abnormal myocardial perfusion | Day 1
  Assess the prevalence of abnormal blood flow in the heart muscle, as defined by a minimum of 2 adjacent cardiac segments each with ≥50% deficit in myocardial perfusion at peak stress revealed by (1) visual assessment of the dynamic stress perfusion CMR scan and (2) pixel mapping of myocardial blood flow (< 2.0 ml/min/g tissue).
Myocardial blood flow | Day 1
  Assess the associations between myocardial blood flow (ml/min/g) and invasive measures of coronary function (where available) that might be implicated in the pathophysiology of abnormal coronary vascular function.
Myocardial tissue characteristics | Day 1
  Assess the correlation between myocardial blood flow (ml/min/g) and myocardial tissue characteristics as revealed by MRI T1- and T2- relaxation times (ms) and extracellular volume fraction.
Cardiovascular risk | Day 1
  Assess the correlation between cardiovascular risk factors, reflected by validated risk scores (e.g. ASSIGN, JBS3), and myocardial blood flow (ml/min/g) in medically managed patients.
Within subject change in myocardial blood flow | 0-12 months
  Assess the within-subject change in cardiac MRI findings during 12-months. This will be done by measuring the within-subject change in peak, global, myocardial blood flow over 12 months.
Between-group, within subject change in myocardial blood flow | 0-12 months
  Assess the between-group, within-subject change in cardiac MRI findings over 12 months. This outcome will provide insights into the effect of the study intervention on MRI findings. This will be done by measuring the within-subject, between group change in peak, global, myocardial blood flow over 12 months.
Health Status: EQ5D-5L Questionnaire | 0-36 months
  The 5-item EuroQol Group EQ5D-5L is a validated questionnaire comprising mobility, self-care, usual activities, pain/discomfort and anxiety/depression to quantitatively assess patient's self-reported health status and will be administered at each study visit.
Health Status: Seattle Angina Questionnaire | 0-36 months
  Seattle Angina Questionnaire (SAQ) Summary Score and component scores (Angina Limitation, Angina Stability, Angina Frequency, Treatment Satisfaction and Quality of Life) will be recorded at all study visits.
Health Status: Illness Perception - Brief IPQ | 0-36 months
  Brief Illness Perception Questionnaire (Brief IPQ), a nine-item scale designed to rapidly assess the cognitive and emotional representations of illness taken at all study visits.
Health Status: Treatment satisfaction - TSQM | 0-36 months
  The 14-item Treatment Satisfaction Questionnaire for Medication (TSQM) is a reliable and valid instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction and will administered at all study visits.
Health Status: Duke Activity Status Index | 0-36 months
  The 12 point Duke Activity Status Index (DASI) is a validated questionnaire to assess functional capacity and will be administered at all study visits.
Health Status: International Physical Activity Questionnaire- Short Form (IPAQ-SF) | 0-36 months
  The 4 point IPAQ-SF is a validated questionnaire to assess functional ability and activuty levels and will be administered at all study visits.
Health Status: Montreal Cognitive Assessment (MOCA) | 0-36 months
  The MOCA is an internationally validated 30 point assessment of cognitive function, and will be administered on all study visits.
Correlation between myocardial blood flow and health status | 0-36 months
  Assess the correlation between myocardial blood flow (ml/min/g) and health status, as measured by validated questionnaires.
Long term prognosis | 0-20 years
  Assess the long-term prognostic significance of between myocardial perfusion (ml/min/g).
Health Outcomes: Major Adverse Cardiovascular Events | 0-20 years
  MACE including death, re-hospitalisation for cardiovascular events including myocardial infarction, heart failure, stroke/ TIA, unstable angina and coronary revascularisation. Unscheduled hospital visits for chest pain that have not led to hospital admission will also be documented.
Angina events | 0-3 years
  Anginal episodes based on completion of a chest symptoms log and adjudicated by a clinical event committee.
Brain small vessel disease | 0-36 months
  Quantify small vessel disease score in the brain using the The STandards for ReportIng Vascular changes on nEuroimaging (STRIVE) guidelines.
Correlation between small vessel disease in the brain and myocardial perfusion | 0-36 months
  Assess the correlation between MRI features of small vessel disease in the brain and myocardial perfusion.
Health economics: Inpatients visits | 0-20 years
  Health resource utilisation will also be assessed by recording the number of inpatient visits in the follow-up period
Health economics: Cardiac procedures | 0-20 years
  Health resource utilisation will also be assessed by recording the number of repeat cardiac procedures performed in the follow up period
Health economics: Medication use | 0-20 years
  Health resource utilisation will also be assessed by recording the medication used in the follow up period
Work limitation | 0-36 months
  Use the 8-item Work limitation Questionnaire to estimate productivity loss and time lost from work, where appropriate.

OTHER OUTCOMES:
Small vessel substudy | 0-12 months
  Sub-study of small vessel function using myography in arterioles isolated from gluteal skin biopsies.
  Standard pharmacological read-outs include the drug concentration required to achieve 50% of the maximum contraction and/or relaxation (wire myography) and structure/function relationships (pressure myography).
Retinal imaging substudy | 0-12 months
  Retinal vascular imaging by optical coherence tomography (OCT) to assess for the presence or absence of small vessel disease.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MBChB, PhD, Principal Investigator — Univerisity of Glasgow
Locations (3):
- United Kingdom (3):
  - University Hospital Hairmyres, East Kilbride, Glasgow
  - University Hospital Ayr, Ayr, Scotland
  - Golden Jubilee National Hospital, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data may be shared based on a research agreement
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the study has completed
Access Criteria: Bone fide collaboration request
URL: http://www.gla.ac.uk/researchinstitutes/icams/staff/colinberry/

REFERENCES:
- [Background] Bradley CP, Berry C. Microvascular arterial disease of the brain and the heart: a shared pathogenesis. QJM. 2023 Oct 23;116(10):829-834. doi: 10.1093/qjmed/hcad158. PMID 37467080
- [Background] Bradley CP, Orchard V, McKinley G, Heggie R, Wu O, Good R, Watkins S, Lindsay M, Eteiba H, McGowan J, McGeoch R, Corcoran D, Kellman P, McConnachie A, Berry C. The coronary microvascular angina cardiovascular magnetic resonance imaging trial: Rationale and design. Am Heart J. 2023 Nov;265:213-224. doi: 10.1016/j.ahj.2023.08.067. Epub 2023 Aug 30. PMID 37657593
- [Background] Bradley C, Berry C. Definition and epidemiology of coronary microvascular disease. J Nucl Cardiol. 2022 Aug;29(4):1763-1775. doi: 10.1007/s12350-022-02974-x. Epub 2022 May 9. PMID 35534718
- [Background] Sidik NP, Stanley B, Sykes R, Morrow AJ, Bradley CP, McDermott M, Ford TJ, Roditi G, Hargreaves A, Stobo D, Adams J, Byrne J, Mahrous A, Young R, Carrick D, McGeoch R, Corcoran D, Lang NN, Heggie R, Wu O, McEntegart MB, McConnachie A, Berry C. Invasive Endotyping in Patients With Angina and No Obstructive Coronary Artery Disease: A Randomized Controlled Trial. Circulation. 2024 Jan 2;149(1):7-23. doi: 10.1161/CIRCULATIONAHA.123.064751. Epub 2023 Oct 5. PMID 37795617
- [Background] Ludman P on behalf of the British Cardiovascular Intervention Society (BCIS). BCIS Audit Returns for Adult Interventional Procedures (Jan - Dec 2016). October 2017. https://www.bcis.org.uk/resources/audit-results/
- [Background] Williams MC, Hunter A, Shah A, Assi V, Lewis S, Mangion K, Berry C, Boon NA, Clark E, Flather M, Forbes J, McLean S, Roditi G, van Beek EJ, Timmis AD, Newby DE; Scottish COmputed Tomography of the HEART (SCOT-HEART) Trial Investigators. Symptoms and quality of life in patients with suspected angina undergoing CT coronary angiography: a randomised controlled trial. Heart. 2017 Jul;103(13):995-1001. doi: 10.1136/heartjnl-2016-310129. Epub 2017 Feb 28. PMID 28246175
- [Background] Ford TJ, Stanley B, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, Sidik N, McCartney P, Corcoran D, Collison D, Rush C, McConnachie A, Touyz RM, Oldroyd KG, Berry C. Stratified Medical Therapy Using Invasive Coronary Function Testing in Angina: The CorMicA Trial. J Am Coll Cardiol. 2018 Dec 11;72(23 Pt A):2841-2855. doi: 10.1016/j.jacc.2018.09.006. Epub 2018 Sep 25. PMID 30266608
- [Background] Ford TJ, Stanley B, Sidik N, Good R, Rocchiccioli P, McEntegart M, Watkins S, Eteiba H, Shaukat A, Lindsay M, Robertson K, Hood S, McGeoch R, McDade R, Yii E, McCartney P, Corcoran D, Collison D, Rush C, Sattar N, McConnachie A, Touyz RM, Oldroyd KG, Berry C. 1-Year Outcomes of Angina Management Guided by Invasive Coronary Function Testing (CorMicA). JACC Cardiovasc Interv. 2020 Jan 13;13(1):33-45. doi: 10.1016/j.jcin.2019.11.001. Epub 2019 Nov 11. PMID 31709984
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Buchanan GL, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. EuroIntervention. 2021 Jan 20;16(13):1049-1069. doi: 10.4244/EIJY20M07_01. PMID 32624456
- [Background] Ford TJ, Berry C. Angina: contemporary diagnosis and management. Heart. 2020 Mar;106(5):387-398. doi: 10.1136/heartjnl-2018-314661. Epub 2020 Feb 12. No abstract available. PMID 32054665
- [Background] Corcoran D, Ford T, Hsu LY, Orchard V, Oldroyd KG, Arai AE, Berry C, on behalf of the CorMicA Investigators. The diagnostic utility of multiparametric CMR in patients with angina and non-obstructive coronary artery disease. Eur Heart J. 2020;
- [Background] Kotecha T, Martinez-Naharro A, Boldrini M, Knight D, Hawkins P, Kalra S, Patel D, Coghlan G, Moon J, Plein S, Lockie T, Rakhit R, Patel N, Xue H, Kellman P, Fontana M. Automated Pixel-Wise Quantitative Myocardial Perfusion Mapping by CMR to Detect Obstructive Coronary Artery Disease and Coronary Microvascular Dysfunction: Validation Against Invasive Coronary Physiology. JACC Cardiovasc Imaging. 2019 Oct;12(10):1958-1969. doi: 10.1016/j.jcmg.2018.12.022. Epub 2019 Feb 13. PMID 30772231
- [Background] Hsu LY, Jacobs M, Benovoy M, Ta AD, Conn HM, Winkler S, Greve AM, Chen MY, Shanbhag SM, Bandettini WP, Arai AE. Diagnostic Performance of Fully Automated Pixel-Wise Quantitative Myocardial Perfusion Imaging by Cardiovascular Magnetic Resonance. JACC Cardiovasc Imaging. 2018 May;11(5):697-707. doi: 10.1016/j.jcmg.2018.01.005. Epub 2018 Feb 14. PMID 29454767
- [Background] Knott KD, Seraphim A, Augusto JB, Xue H, Chacko L, Aung N, Petersen SE, Cooper JA, Manisty C, Bhuva AN, Kotecha T, Bourantas CV, Davies RH, Brown LAE, Plein S, Fontana M, Kellman P, Moon JC. The Prognostic Significance of Quantitative Myocardial Perfusion: An Artificial Intelligence-Based Approach Using Perfusion Mapping. Circulation. 2020 Apr 21;141(16):1282-1291. doi: 10.1161/CIRCULATIONAHA.119.044666. Epub 2020 Feb 14. PMID 32078380
- [Background] Berry C, Sidik N, Pereira AC, Ford TJ, Touyz RM, Kaski JC, Hainsworth AH. Small-Vessel Disease in the Heart and Brain: Current Knowledge, Unmet Therapeutic Need, and Future Directions. J Am Heart Assoc. 2019 Feb 5;8(3):e011104. doi: 10.1161/JAHA.118.011104. No abstract available. PMID 30712442
- [Background] Ford TJ, Rocchiccioli P, Good R, McEntegart M, Eteiba H, Watkins S, Shaukat A, Lindsay M, Robertson K, Hood S, Yii E, Sidik N, Harvey A, Montezano AC, Beattie E, Haddow L, Oldroyd KG, Touyz RM, Berry C. Systemic microvascular dysfunction in microvascular and vasospastic angina. Eur Heart J. 2018 Dec 7;39(46):4086-4097. doi: 10.1093/eurheartj/ehy529. PMID 30165438
- [Derived] Bradley CP, McKinley G, Orchard V, Tiller C, Stanley B, Ang D, Morrow AJ, Sykes R, Gildea P, Petty M, Brogan R, Carrick D, Collison D, Eteiba H, Ghattas A, Good R, Joshi F, Lindsay M, McCartney P, McGowan J, McGeoch R, Robertson K, Rocchiccioli P, Shaukat A, Watkins S, Kellman P, McConnachie A, Berry C. Endotyping-informed therapy for patients with chest pain and no obstructive coronary artery disease: a randomized trial. Nat Med. 2026 Jan;32(1):332-341. doi: 10.1038/s41591-025-04044-4. Epub 2025 Nov 10. PMID 41214345
- [Derived] Bradley CP, Orchard V, Sykes RA, McKinley G, McConnachie A, Donnelly P, Watt J, Kellman P, Quinn T, Fullerton N, Berry C. Heart-brain microvascular MRI study: protocol for a multicentre, observational, cohort study in the UK assessing associations between small vessel disease of the heart and brain. BMJ Open. 2024 Dec 20;14(12):e088372. doi: 10.1136/bmjopen-2024-088372. PMID 39806582